CLINICAL TRIAL: NCT05405114
Title: A Multicentre Trial Evaluating the Efficacy and Safety of Oral Decitabine Tetrahydrouridine (NDec) in Patients With Sickle Cell Disease
Brief Title: Research Study Investigating How Well NDec Works in People With Sickle Cell Disease
Acronym: ASCENT1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN7533-4470; U1111-1255-1324 (Other: World Health Organization (WHO)); 2020-003485-39 (EudraCT Number)
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- HU-non-eligible - NDec plus placebo (Experimental): HU-non eligible patients randomised to treatment with NDec on one day and placebo on the other day
  Interventions: Drug: NDec - oral decitabine-tetrahydrouridine; Drug: Placebo
- HU-non-eligible - NDec plus NDec (Experimental): HU-non eligible patients randomised to treatment with NDec on both days
  Interventions: Drug: NDec - oral decitabine-tetrahydrouridine
- HU-non-eligible - Placebo plus placebo (Placebo Comparator): HU-non eligible patients randomised to treatment with placebo on both days
  Interventions: Drug: Placebo
- HU-active - NDec plus placebo (Experimental): HU-active patients randomised to treatment with NDec on one day and placebo on the other day
  Interventions: Drug: NDec - oral decitabine-tetrahydrouridine; Drug: Placebo
- HU-active - NDec plus NDec (Experimental): HU-active patients randomised to treatment with NDec on both days
  Interventions: Drug: NDec - oral decitabine-tetrahydrouridine
- HU-active - HU (Active Comparator): HU-active patients randomised to continue on open-label HU treatment
  Interventions: Drug: HU - Hydroxyurea

INTERVENTIONS:
Drug: NDec - oral decitabine-tetrahydrouridine — Participants will get capsules (oral administration) to take once or twice weekly. The number of capsules will be based on their body weight
  Arms: HU-active - NDec plus NDec; HU-active - NDec plus placebo; HU-non-eligible - NDec plus NDec; HU-non-eligible - NDec plus placebo
Drug: HU - Hydroxyurea — Participants will get capsules daily (oral administration) according to local labelling
  Arms: HU-active - HU
Drug: Placebo — Participants will get capsules (oral administration) to take once or twice weekly. The number of capsules will be based on their body weight
  Arms: HU-active - NDec plus placebo; HU-non-eligible - NDec plus placebo; HU-non-eligible - Placebo plus placebo

SUMMARY:
This study examines how well a new, potential medicine called NDec works and is tolerated in people with sickle cell disease. NDec is a combination of two medicines (decitabine-tetrahydrouridine). Both medicines are new for the treatment of sickle cell disease. Participants who are not taking Hydroxyurea (HU) will get NDec, NDec and placebo, or placebo. Participants who are on HU treatment before joining the study will get NDec, NDec and placebo, or continue on HU. Which treatment participants get is decided by chance. Participants getting NDec and/or Placebo will get capsules to take twice weekly. The study will last for about a year.

ELIGIBILITY:
Inclusion Criteria:

* Age above or equal to 18 years at the time of signing informed consent
* Confirmed diagnosis of SCD (including HbSS, HbSC, HbSβ0 thalassaemia and HbSβ+ thalassaemia or other Sickle Cell disease variants)
* 2-10 episodes of documented vaso-occlusive crisis (VOCs) within the last 12 months prior to the screening visit
* Haemoglobin greater than or equal to 5.0 g/dL and below or equal to 10.5 g/dL at visit 1
* Absolute reticulocyte count above upper limit of the normal (ULN) at visit 1
* Body weight 40 to 125 kg (inclusive).

Exclusion Criteria:

* Patient is on chronic transfusion therapy as defined by receiving scheduled (pre-planned) series of blood transfusion (simple or exchange) for prophylactic purposes, or the patient is likely to begin chronic transfusion therapy during the course of the trial, or has received RBC or whole blood transfusion for any reason within 28 days of visit 1
* Receipt of erythropoietin or other haematopoietic growth factor treatment within 28 days of signing ICF, or planned treatment with these agents during the trial
* Receipt of voxelotor, crizanlizumab or L-glutamine treatment within 12 weeks of signing the informed consent form, or planned treatment with such agents during the trial
* Platelet count greater than 800 x 10^9/L at visit 1
* Absolute neutrophil count below or equal to 1.5 x 10^9/L at visit 1
* Any condition/concurrent chronic disease involving the stomach or small intestine which may affect drug absorption, as per investigator's judgement
* Female who is

  * pregnant, breast-feeding or intends to become pregnant within 6 months after the final trial product administration
  * child-bearing potential and not using highly effective methods of contraception and whose male partner is not using effective contraception, at screening and until 6 months after the last dose of trial product
* Male with female partner of childbearing potential who does not agree to use condom and whose female partner of childbearing potential is not using a highly effective contraceptive measure from trial start to:

  * Six (6) months after the last dose of trial product for patients on NDec/Placebo
  * Six (6) months after the last dose of trial product for patients outside US and CA randomised to HU
  * Twelve (12) months after the last dose of trial product for patients randomised to HU in US and CA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Change in total haemoglobin | From baseline (week 0) to week 24
  measured in g/dL

SECONDARY OUTCOMES:
Cmax for decitabine from pharmacokinetic assessment | At week 24
  measured in ng/mL
Cmax for tetrahydrouridine from pharmacokinetic assessment | At week 24
  measured in ng/mL
Change in DNA methyltransferase 1 (DNMT1) activity | From baseline (week 0) to week 24
  measured in MFI units
Change in cytidine deaminase (CDA) activity | From baseline (week 0) to week 24
  µmol/L/min
Change in foetal haemoglobin (g/dL) | From baseline (week 0) to week 24
  measured in g/dL
Change in foetal haemoglobin as a proportion of total haemoglobin (%HbF) | From baseline (week 0) to week 24
  measured in %
Change in F-cell level as a proportion of total red blood cell (RBC) (%F-cells) | From baseline (week 0) to week 24
  measured in %
Change in haemolysis measure: absolute reticulocyte count | From baseline (week 0) to week 24
  measured in cells × 10^9/L
Change in haemolysis measure: indirect bilirubin | From baseline (week 0) to week 24
  measured in mg/dL
Change in haemolysis measure: lactate dehydrogenase | From baseline (week 0) to week 24
  measured in U/L
Number of vaso-occlusive crises | From baseline (week 0) to week 48
  number of events
Number of acute chest syndrome | From baseline (week 0) to week 48
  number of events
Number of RBC units transfused | From baseline (week 0) to week 48
  measured in Units
Number of adverse events of grade 3 or higher | From baseline (week 0) to week 52
  number of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (65):
- United States (20):
  - University Of South Alabama, Mobile, Alabama
  - UCSF Oakland Benioff Children's Hospital, Oakland, California
  - Center for Inherited Blood Dis, Orange, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Clinical and Transl Res Center, Aurora, Colorado
  - Howard University, Washington D.C., District of Columbia
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - University of Miami Hospital & Clinics, Miami, Florida
  - University Of Illinois at Chicago, Chicago, Illinois
  - Tulane Sickle Cell Ctr- So LA, Metairie, Louisiana
  - Mississippi Center Advanced Medicine, Madison, Mississippi
  - Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Mount Sinai School of Medicine, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - East Carolina Univ-Greenville, Greenville, North Carolina
  - Univ Oklahoma HSC_Okla City, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center_Oklahoma City, Oklahoma City, Oklahoma
  - St Christopher Hosp for Child, Philadelphia, Pennsylvania
  - Medical Univ of SC Charleston, Charleston, South Carolina
  - Univ Texas HSC-Houston, Houston, Texas
- Canada (3):
  - LHSC - Victoria Hospital, London, Ontario
  - Toronto General Hospital, Liver Clinic, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- France (2):
  - Centre Hospitalier Universitaire Grenoble Alpes-Site Nord Michallon-3, Grenoble
  - Hospices Civils de Lyon-Hopital Edouard Herriot, Lyon
- Greece (3):
  - Aghia Sophia Childrens' Hospital, Goudi
  - General Hospital Of Larissa Koutlibaneio And Triantafylleio - Thalassemia and SCD Unit, Larissa
  - Gen Univ Hospital of Patras, Thalassemia/Hemoglobinopathies, Pátrai
- India (18):
  - All India Institute of Medical Sciences (AIIMS), Raipur, Raipur, Chhattisgarh
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - BAPS Pramukh Swami Hospital, Surat, Gujarat
  - SSG Hospital, Baroda, Vadodara, Gujarat
  - Victoria Hospital (Bangalore Medical College and Research Institute), Bangalore, Karnataka
  - J.S.S.Hospital, Mysore, Karnataka
  - Government Medical College, Kozhikode, Kozhikode, Kerala
  - K.J Somaiya Hospital and Research Centre, Mumbai, Maharashtra
  - Government Medical College and Hospital, Nagpur, Maharashtra
  - Government Medical College and Super Speciality Hospital, Nagpur, Nagpur, Maharashtra
  - IMS and SUM Hospital, Bhubaneswar, Odisha
  - S.C.B. Medical College, Cuttack, Odisha
  - Christian Medical College Hospital, Vellore, Ranipet, Tamil Nadu
  - Christian Medical College Hospital, Vellore, Vellore, Tamil Nadu
  - Yashoda hospital, Hyderabad, Telangana
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - NRS Medical College & Hospital, Kolkata, West Bengal
  - KIMS - Kingsway Hospital, Nagpur
- Italy (5):
  - Ospedali Galliera, Genova
  - Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedale Universita Padova, Padua
  - Azienda Ospedaliera Universitaria Integrata Verona Policlinico GB Rossi - Borgo Roma, Verona
  - Policlinico GB Rossi, Verona
- Hospital Nini, Tripoli, Lebanon
- Sultan Qaboos University Hospital, Muscat, Oman
- Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Johannesburg, Gauteng, South Africa
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- Turkey (Türkiye) (4):
  - Acıbadem Adana Hastanesi-Hematoloji, Adana
  - Çukurova Üniversitesi Tıp Fakültesi Balcalı Hastanesi- Hematoloji, Adana
  - Hacettepe Üniversitesi Hastanesi- Hematoloji, Ankara
  - Mersin Üniversitesi Tip Fakültesi Hastanesi- Çiftlikköy Yerleşkesi- Hematoloji, Mersin
- United Kingdom (5):
  - University Hospital of Wales, Cardiff
  - Central Middlesex Hospital, London
  - Guy's Hosptial, London
  - Kings College Hospital, London
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Helleberg H, Bjornsdottir I, Offenberg HK. Effects of Tetrahydrouridine Pre-dosing on Absorption, Metabolism, and Excretion of Decitabine in the Mouse. Eur J Pharm Sci. 2026 Jan 1;216:107353. doi: 10.1016/j.ejps.2025.107353. Epub 2025 Oct 27. PMID 41161613
- [Derived] Abbasi M, Srivastava A, Saraf SL. Management of Kidney Disease with Sickle Cell Disease. J Am Soc Nephrol. 2025 Oct 1;36(10):2041-2054. doi: 10.1681/ASN.0000000804. Epub 2025 Jun 26. PMID 40569673